CLINICAL TRIAL: NCT05669508
Title: The Reynolds Innovative Spinal Electrical Stimulation (RISES) Program: Transcutaneous Spinal Cord Stimulation
Brief Title: Wearable Electrical Stimulation on the Back to Modulate Spinal Cord Activity
Acronym: RISES-T
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Mijail Demian Serruya, Assistant Professor, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Rises-T 22D.126
Record Dates: First submitted 2022-11-16; First posted 2023-01-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
Keywords: Spinal Cord Injuries; Spinal Electrical Stimulation; Transcutaneous Spinal Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Participants will receive closed-loop transcutaneous spinal cord stimulation via the RISES-T System while completing functional task practice in occupational therapy sessions.
  Interventions: Device: RISES-T System; Other: Occupational/Physical Therapy

INTERVENTIONS:
Device: RISES-T System — Non-invasive closed-loop electrical stimulation of the spinal cord through the skin
  Other Names: Transcutaneous spinal stimulation
Other: Occupational/Physical Therapy — Exercise therapy to improve function of upper and/or lower limbs
  Other Names: Functional Task Practice

SUMMARY:
The goal of this study is to evaluate if non-invasive electrical spinal stimulation can help people with paralysis caused by SCI improve strength and function of their arms, legs, hands or feet. The study will involve therapy sessions involving exercises done at the same time as electrical stimulation therapy. This study has multiple parts to evaluate the effectiveness and safety of "smart" electrical stimulation of the spinal cord, which involves stimulating the spinal cord at precise locations and times to improve movement and function.

DETAILED DESCRIPTION:
This trial is investigating the use of transcutaneous spinal cord stimulation, where the electrical stimulation is delivered non-invasively via surface electrodes placed on the skin along the spine. The trial will have two phases: open-loop transcutaneous spinal cord stimulation (SCS) phase (where stimulation parameters are selected and subsequently fixed for each stimulation sessions) and closed-loop transcutaneous SCS phase, (where stimulation parameters are continuously revised in real-time during each session based upon the exact movement state of the person as captured by wearable kinematic and electromyographic sensors). For both open-loop and closed-loop phases, the transcutaneous spinal cord stimulation will be incorporated into Functional Task Practice (FTP) sessions guided closely by a team of trained technicians and occupational and physical therapists.

Upon enrollment, participants will complete a baseline assessment of outcome measures validated for spinal cord injury rehabilitation. They will also undergo mapping with sensors of their movements without stimulation to simply characterize their unique "motor signature". Then they will undergo the same mapping with open-loop transcutaneous SCS applied to determine if and how stimulation at a variety of settings can modify their unique "motor signature". They will then participate in the open-loop phase - 15 open-loop SCS+FTP sessions - after which they will repeat the outcome measures (interim assessment). They will then proceed to the closed-loop phase - 15 closed-loop SCS+FTP sessions - after which they will repeat the outcome measures a final time (endpoint assessment).

ELIGIBILITY:
Inclusion Criteria:

* Has a non-progressive or central cord spinal cord injury from C2-T10 inclusive
* Has American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification B, C, or D
* Can participate in physical and occupational therapy rehabilitation programs
* Is at minimum 12 months post- spinal cord injury
* Can provide informed consent
* Has adequate caregiver support to facilitate participation in study

Exclusion Criteria:

* Has uncontrolled cardiopulmonary disease or cardiac symptoms (as determined by the Investigator)
* Has diffuse lower motor neuron injury rendering majority of muscles not excitable
* Has any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations like severe neuropathic pain, depression, mood disorders or other cognitive disorders
* Has autonomic dysreflexia that is severe, unstable, and uncontrolled or uncontrolled orthostatic hypotension that may interfere with rehabilitation.
* Requires ventilator support
* Has an autoimmune etiology of spinal cord dysfunction/injury
* Has spasms that limit the ability to participate in the study training (as determined by the Investigator)
* Has skin breakdown in area(s) that will come into contact with electrodes
* Has any active implanted medical device
* Is pregnant, planning to become pregnant or currently breastfeeding
* Has concurrent participation in another drug or device trial that may interfere with this study
* Has other traumatic injuries such as peripheral nerve injuries, severe musculoskeletal injuries (e.g., shattered pelvis, long bone fractures), that prevent evaluation of response to or participation in rehabilitation.
* Is deemed ineligible because the investigators believe the study would not be safe or appropriate for the individual

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline- International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | Repeated measurements once every 6 weeks throughout the study, an average of 3 months
  Standard neurological assessment for determining level and severity of impairment after spinal cord injury. It includes a sensory exam (dermatological light touch and pin prick) and motor exam (manual muscle strength testing).

SECONDARY OUTCOMES:
Change from Baseline - Spinal Cord Independence Measures (SCIM) | Repeated measurements once every 6 weeks throughout the study, an average of 3 months
  Validated measure that evaluates self-care (feeding, grooming, bathing, dressing), respiration and sphincter management, and mobility abilities (transfers and indoor/outdoor).
Change from Baseline - Canadian Occupational Performance Measure (COPM) | Repeated measurements once every 6 weeks throughout the study, an average of 3 months
  Participant-centered instrument that measures changes in how participants perceive their own functional performance and challenges in daily living; participants identify goals of most importance to them in areas of functional tasks and occupational performance including self-care, leisure, and productivity.
Change from Baseline - Capabilities of Upper Extremity (CUE-T) | Repeated measurements once every 6 weeks throughout the study, an average of 3 months
  Validated objective measure of upper extremity functional capabilities in persons with SCI; evaluates the ability to perform various actions (reach up, pull up, picking up a pencil with tips of fingers).
Change from 10 Meter Walk Test (10MWT) and Walking Index for Spinal Cord Injury (WISCI II) | Repeated measurements once every 6 weeks throughout the study, an average of 3 months
  Validated performance measures to assess walking speed and amount of physical assistance needed/assistive devices required for walking respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mijail D Serruya, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Background] Manson G, Atkinson DA, Shi Z, Sheynin J, Karmonik C, Markley RL, Sayenko DG. Transcutaneous spinal stimulation alters cortical and subcortical activation patterns during mimicked-standing: A proof-of-concept fMRI study. Neuroimage Rep. 2022 Jun;2(2):100090. doi: 10.1016/j.ynirp.2022.100090. Epub 2022 Mar 8. PMID 36212800
- [Background] Kumru H, Rodriguez-Canon M, Edgerton VR, Garcia L, Flores A, Soriano I, Opisso E, Gerasimenko Y, Navarro X, Garcia-Alias G, Vidal J. Transcutaneous Electrical Neuromodulation of the Cervical Spinal Cord Depends Both on the Stimulation Intensity and the Degree of Voluntary Activity for Training. A Pilot Study. J Clin Med. 2021 Jul 25;10(15):3278. doi: 10.3390/jcm10153278. PMID 34362062
- [Background] Rejc E, Smith AC, Weber KA 2nd, Ugiliweneza B, Bert RJ, Negahdar M, Boakye M, Harkema SJ, Angeli CA. Spinal Cord Imaging Markers and Recovery of Volitional Leg Movement With Spinal Cord Epidural Stimulation in Individuals With Clinically Motor Complete Spinal Cord Injury. Front Syst Neurosci. 2020 Oct 21;14:559313. doi: 10.3389/fnsys.2020.559313. eCollection 2020. PMID 33192348
- [Background] Barss TS, Parhizi B, Porter J, Mushahwar VK. Neural Substrates of Transcutaneous Spinal Cord Stimulation: Neuromodulation across Multiple Segments of the Spinal Cord. J Clin Med. 2022 Jan 27;11(3):639. doi: 10.3390/jcm11030639. PMID 35160091
- [Background] Capogrosso M, Wagner FB, Gandar J, Moraud EM, Wenger N, Milekovic T, Shkorbatova P, Pavlova N, Musienko P, Bezard E, Bloch J, Courtine G. Configuration of electrical spinal cord stimulation through real-time processing of gait kinematics. Nat Protoc. 2018 Sep;13(9):2031-2061. doi: 10.1038/s41596-018-0030-9. PMID 30190556
- [Background] Wenger N, Moraud EM, Gandar J, Musienko P, Capogrosso M, Baud L, Le Goff CG, Barraud Q, Pavlova N, Dominici N, Minev IR, Asboth L, Hirsch A, Duis S, Kreider J, Mortera A, Haverbeck O, Kraus S, Schmitz F, DiGiovanna J, van den Brand R, Bloch J, Detemple P, Lacour SP, Bezard E, Micera S, Courtine G. Spatiotemporal neuromodulation therapies engaging muscle synergies improve motor control after spinal cord injury. Nat Med. 2016 Feb;22(2):138-45. doi: 10.1038/nm.4025. Epub 2016 Jan 18. PMID 26779815
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197